CLINICAL TRIAL: NCT07379710
Title: Concomitant Use of Norepinephrine With Ephedrine Versus Norepinephrine Alone to Maintain Arterial Blood Pressure During Spinal Anesthesia for Cesarean Delivery, a A Prospective Double-blinded Study.
Brief Title: Norepinephrine With Ephedrine Versus Norepinephrine Alone During Spinal Anesthesia for Cesarean Delivery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Youssef, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS-528-2023
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Incidence of Post-spinal Hypotension
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group(A) (Active Comparator): Ephedrine 10 mg (2.5mg/ml) direct I.V will be given simultaneous with Norepinephrine infusion 0.08 mcg/kg/min
  Interventions: Drug: Ephedrine and Norepinephrine infusion
- Group (B) (Active Comparator): 4 ml normal saline direct I.V will be given simultaneous with norepinephrine (to keep blinding) Infusion 0.08 mcg/kg/min only be infused
  Interventions: Drug: Norepinephrine infusion

INTERVENTIONS:
Drug: Ephedrine and Norepinephrine infusion — Ephedrine 10 mg (2.5mg/ml) direct I.V will be given simultaneous with Norepinephrine infusion 0.08 mcg/kg/min
  Arms: Group(A)
Drug: Norepinephrine infusion — 4 ml normal saline direct I.V will be given simultaneous with norepinephrine (to keep blinding) Infusion 0.08 mcg/kg/min only be infused
  Arms: Group (B)

SUMMARY:
We hypothesize that the addition of ephedrine to norepinephrine infusion could decrease the incidence of post spinal hypotension(PSH) in parturient undergoing C.S under spinal anesthesia and minimize the changes in heart rate

DETAILED DESCRIPTION:
Aim of the work: To compare between concomitant use of norepinephrine infusion with ephedrine versus use of norepinephrine infusion alone on maternal B.P following induction of spinal anaesthesia for C.S delivery.

Statistical analysis Sample Size: Our primary outcome is the incidence of post-spinal hypotension. In a previous study incidence of post spinal hypotension in the noradrenaline group was 32%. We calculated a sample size that could detect at least 50% difference between study groups. Using MedCalc Software version 14 (MedCalc Software bvba, Ostend, Belgium), a sample size of 246 patients will be needed to have a study power of 80% and alpha error of 0.05. The number was increased to be 260 envelopes (130 envelopes per group) to compensate for possible dropouts.

Statistical analysis:

Analysis of data will be performed using Statistical package for social science (SPSS) software, version 26 for Microsoft Windows (SPSS Inc., Chicago, iL, USA). Categorical data will be reported as frequency and percentages and will be analyzed using chi-squared test. Continuous data will be checked for normality using Kolmogorov-Smirnov test. Normally distributed data will be presented as means ±standard deviations and will be analyzed using unpaired student t-test.

Skewed data will be expressed as medians(quartiles) and will be analyzed using Mann Whitney U test. A two-way repeated measures ANOVA will be used to evaluate dose (between-groups factor) and time (repeated measures)". P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II
* Age: 18 to 40 years
* Undergoing Elective Lower Segment Cesarean Section under Spinal Anesthesia.

Exclusion Criteria:

* Uncontrolled cardiac morbidities As reduction of ejection fraction< 60%, History (within 3months) of myocardial infarction, cerebrovascular accident, transient ischemic attacks or coronary artery disease/stents
* Poorly controlled Hypertensive disorders of pregnancy
* Peripartum bleeding
* Coagulation disorders
* Baseline systolic blood pressure (SBP) < 100 mmHg
* Refusal of patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-spinal hypotension | Baseline (T0), just after spinal anaesthesia (T1) then every 2.5 minutes until delivery of the fetus

SECONDARY OUTCOMES:
Incidence of bradycardia | Baseline (T0), just after spinal anaesthesia (T1) then every 2.5 minutes until delivery of the fetus
  Defined as heart rate < 55 bpm
Reactive hypertension | Baseline (T0), just after spinal anaesthesia (T1) then every 2.5 minutes until delivery of the fetus
  Defined as SBP > 120% from the baseline reading
Systolic blood pressure | Baseline (T0), just after spinal anaesthesia (T1) then every 2.5 minutes until delivery of the fetus
Heart rate | Baseline (T0), just after spinal anaesthesia (T1) then every 2.5 minutes until delivery of the fetus
Rescue vasopressor consumption | Just after spinal anaesthesia until delivery of the fetus
  Cumulative intraoperative boluses of ephedrine and norepinephrine doses
Neonatal outcomes Apgar Score | Within 5 minutes of baby delivery
  The Apgar score comprises five components: 1- color, 2- heart rate, 3- reflexes, 4- muscle tone, and 5- respiration, each of which is given a score of 0, 1, or 2

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ollaek, MD, Principal Investigator — Faculty of Medicine, Cairo University, Cairo
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No